CLINICAL TRIAL: NCT07292714
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Study to Evaluate Efficacy and Safety of 9MW1911 in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Study to Evaluate 9MW1911 in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9MW1911-2025-CP201
Record Dates: First submitted 2025-12-02; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Chronic Obstructive Pulmonary Disease COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase II 9MW1911 (Experimental): 9MW1911 is administered intravenously in two dose levels. Each dose group include 120 patients.
  Interventions: Drug: 9MW1911
- Phase II Placebo (Placebo Comparator): Phase II Placebo is administered intravenously. this group includes 120 patients.
  Interventions: Drug: Phase II placebo

INTERVENTIONS:
Drug: 9MW1911 — Participants will receive IV 9MW1911 in each dose every 28 days.
  Arms: Phase II 9MW1911
Drug: Phase II placebo — Participants will receive IV placebo every 28 days.
  Arms: Phase II Placebo

SUMMARY:
The study is a Phase II, multicenter, double-blind, randomized, parallel, placebo-controlled clinical trial designed to evaluate the efficacy, safety of 9MW1911 in patients with Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

- 1.Male or Female patients must be 40 to 75 years of age inclusive； 2.Physician diagnosis of COPD for at least 1 year at screening； 3.Documented history of >= 2 moderate or >=1 severe COPD exacerbations within 12 months prior to screening.

4.Moderate-to-severe COPD with post-BD FEV1/FVC rato<0.7 and a post-BD FEV1%predicted ≥20% and<80% at screening； 5.Body Mass Index (BMI) of 16 kg/m² to 32 kg/m²； 6.Current tobacco smoker or former smoker with a history of smoking ≥ 10 pack-years 7.Participants with standard of care controller therapy, for ≥3 months prior to Screening and at a stable dose of controller therapy for at least 1 month prior to the screening；

Exclusion Criteria:

* 1.Current diagnosis of asthma or documented history of asthma; 2.Diagnosis of Alpha-1 Antitrypsin Deficiency； 3.History of other clinically significant pulmonary diseases apart from COPD: such as sarcoidosis,interstitial lung diseases, bronchiectasis,cystic fibrosis，constrictive bronchiolitis,severe pulmonary hypertension or other active pulmonary diseases; 4.Long-term treatment with oxygen (oxygen therapy time >15h/day) or mechanical ventilation, or clinically significant apnea requiring continuous positive airway pressure (CPAP) or non-invasive positive pressure ventilation (NIPPV); 5.History of lung pneumonectomy, or lung volume reduction within 12 months prior to screening，or planned to undergo lung volume reduction surgery (LVRS) during the study period; 6.Patients in the acute phase of pulmonary rehabilitation(participating in, or scheduled for a pulmonary rehabilitation program within 4 weeks of screening); 7.Uncured upper or lower respiratory tract infections during the screening period; 8.Moderate to severe COPD exacerbations within 4 weeks prior to screening or during the screening period； 9.Any infection requiring hospitalization for ≥24 hours and/or treatment with oral, IV, or IM antibiotics within 4 weeks prior to screening or during the screening period; 10.Received treatment with oral, IV, or intramuscular (IM) corticosteroids (>10 mg/day prednisone or equivalent dose) within 4 weeks prior to starting study medication; 11.Myocardial infarction, unstable angina within 12 months prior to screening;or heart failure (NYHA Class III or IV) within 6 months prior to screening； 12.History of ventricular arrhythmias or risk factors for ventricular arrhythmias, such as structural heart disease (e.g., severe left ventricular systolic dysfunction, severe left ventricular hypertrophy ), family history of unexplained sudden death or long QT syndrome； 13. experienced transient ischemic attack or stroke within 6 months prior to screening; 14.with unstable cardiovascular diseases, such as pulmonary embolism or deep vein thrombosis that occurred within 6 months before screening, which the researchers believe may put the patient at risk or have a negative impact on the research results; 15.Known active tuberculosis or nontuberculous mycobacterial infection (subjects with positive interferon - γ release assay (IGRA) during the screening period, if evaluated as inactive tuberculosis by the researcher based on clinical manifestations and imaging examinations, etc., can participate in this study); 16.Positive for human immunodeficiency virus antibody (HIV-Ab), or positive for hepatitis B surface antigen (HBsAg) with HBV-DNA copies > 1000 IU/mL or above the upper limit of normal (ULN) of the study center, or positive for hepatitis C virus antibody (HCV-Ab) with HCV-RNA copies above the ULN of the study center, or positive for Treponema pallidum antibody.

  17.With active autoimmune disease or receiving immunosuppressive therapy for an autoimmune diseases (e.g., rheumatoid arthritis, inflammatory bowel disease, primary biliary cirrhosis, systemic lupus erythematosus, multiple sclerosis) are excluded.

  18. with any active malignancy or a history of malignancy (except for low-grade tumors deemed cured ≥5 years before screening, such as cervical carcinoma in situ or basal cell carcinoma).

  19.received a live attenuated vaccine within 4 weeks prior to screening or during the screening period.

  20.received any biologic therapy (e.g., omalizumab, dupilumab, and/or anti-interleukin-5 therapy) within 3 months prior to screening ; 21.received any investigational therapy within 3 months prior to screening or within 5 drug-elimination half-lives, whichever is longer.

  22.Any clinically significant ECG abnormality deemed by the investigator to potentially affect study conduct, such as QTc prolongation (QTcF > 450 ms for males, > 470 ms for females).

  23.Alanine aminotransferase (ALT) >= 2 times the upper limit of normal (ULN); Aspartate aminotransferase (AST) >= 2 times ULN; Total bilirubin >= 1.5 times ULN.

  24.Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2. 25.with any serious medical condition or clinically significant laboratory abnormality（in investigator's judgment） that could compromise the subject's safety or ability to participate in or complete the study.

  26. With a history of alcohol abuse and/or substance abuse within 12 months prior to screening.

  27.History of severe hypersensitivity or anaphylactic reactions to any biologic agent, or known hypersensitivity to any component of the investigational drug.

  28. Pregnant or lactating women, Or female paticipants of child-bearing potential with a positive pregnancy test at screening.

  29.Subjects who is inappropriate to participate in the trial due to any reasons as determined by the investigator.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
The annualized incidence rate of moderate to severe acute exacerbations of chronic obstructive pulmonary disease (AECOPD） within 52 weeks | Baseline up to week 52
  Within a 52-week period, the number of acute exacerbations of chronic obstructive pulmonary disease (AECOPD) is converted to an annual incidence rate.

SECONDARY OUTCOMES:
Changes from baseline in pre-bronchodilator FEV1 | Weeks 0, 4, 8, 12,24,36,52
  Changes in pre-bronchodilator FEV1 levels at 4, 8, 12, 24，36 and 52 weeks compared to baseline.
Changes from baseline in post-bronchodilator FEV1 | Weeks 0, 4, 8, 12,24,36,52
  Changes in post-bronchodilator FEV1 levels at 4, 8, 12, 24，36and 52 weeks compared to baseline.
Changes from baseline in pre-bronchodilator FVC | Weeks 0, 4, 8, 12,24,36,52
  Changes in pre-brochodilator FVC levels at 4, 8, 12, 24，36 and 52 weeks compared to baseline.
Changes from baseline in post-bronchodilator FVC | Weeks 0, 4, 8, 12,24,36,52
  Changes in post-bronchodilator FVC levels at 4, 8, 12, 24，36 and 52 weeks compared to baseline.
Time to first moderate to severe Chronic Obstructive Pulmonary Disease Acute Exacerbation (AECOPD) from baseline to week 52. | Baseline to week 52
  Time to first moderate to severe Chronic Obstructive Pulmonary Disease Acute Exacerbation (AECOPD) from baseline to week 52.
Annualized rate of moderate to severe AECOPD over the 52-week treatment period. | Baseline to week 52
  Within a 52-week period, the number of severe acute exacerbations of chronic obstructive pulmonary disease (AECOPD) is converted to an annual incidence rate.
Time to first severe Chronic Obstructive Pulmonary Disease Acute Exacerbation (AECOPD) from baseline to week 52. | Baseline up to week 52
  Time to first severe Chronic Obstructive Pulmonary Disease Acute Exacerbation (AECOPD) from baseline to week 52.
The change from baseline in the St. George's Respiratory Questionnaire-COPD (SGRQ-C) total score | Weeks 0, 4, 12, 24,36,52
  Changes in St. George's Respiratory Questionnaire-COPD (SGRQ-C) total score at 4, 12, 24，36 and 52 weeks compared to baseline.
The proportion of subjects with a ≥4-point improvement from baseline in the total score of the St. George's Respiratory Questionnaire for COPD (SGRQ-C) at Weeks 4, 12, 24, 36, and 52 | Weeks 0, 4, 12, 24,36,52
  The proportion of subjects achieving improvement of ≥4 points from baseline in the St. George's Respiratory Questionnaire for COPD (SGRQ-C) total score at Weeks 4, 12, 24, 36, and 52.
Changes from baseline in CAT(COPD Assessment Test) score at 4，12 ，24，36 and 52 weeks. | Weeks 0, 4, 12, 24，36，52
  Changes in CAT score at 4，12，24，36 and 52 weeks compared to baseline.
Safety and tolerability assessment | 60 weeks
  The incidence and severity of adverse events, adverse reactions, serious adverse events, as well as abnormal clinical laboratory test indicators, vital signs, physical examinations, and 12-lead electrocardiograms.
Immunogenicity Assessment | 52 weeks
  The incidence of Anti-Drug Antibodies (ADA) and Neutralizing Antibodies (Nab).
serum concentrations of 9MW1911 | 32 weeks
  Pharmacokinetics: concentrations of 9MW1911 in serum.
Biological Marker | 52 weeks
  Serum levels of IL-33, IL-5, IL-13, and total sST2, and phosphorylated P38 (p-P38) .
Pharmacogenomics Characteristics | week 0
  Single nucleotide polymorphism of gene rs10206753

CONTACTS AND LOCATIONS:
Locations (51):
- China (51):
  - Chizhou Central Hospital, Chizhou, Anhui
  - Anhui Chest Hospital, Hefei, Anhui
  - Gansu Provincial People's Hospital, Lanzhou, Gansu
  - Huizhou Third People's Hospital, Huizhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Qingyuan Hospital Affiliated to Guangzhou Medical University, Qingyuan, Guangdong
  - The Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Hebei PetroChina Central Hospital, Langfang, Hebei
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Xinxiang First People's Hospital, Xinxiang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Jingzhou First People's Hospital, Jinzhou, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - The Third Hospital of Changsha, Changsha, Hunan
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - Shaoyang Central Hospital, Shaoyang, Hunan
  - Xiangyang Central Hospital, Xiangyang, Hunan
  - Yongzhou Central Hospital, Yongzhou, Hunan
  - Yueyang Central Hospital, Yueyang, Hunan
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Jiujiang First People's Hospital, Jiujiang, Jiangxi
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Inner Mongolia Baogang Hospital, Baotou, Neimenggu
  - Heze Municipal Hospital, Heze, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shandong Provincial Public Health Clinical Center, Jinan, Shandong
  - Weifang Second People's Hospital, Weifang, Shandong
  - Jinmei Group General Hospital, Jincheng, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Xi'an Chest Hospital, Xi’an, Shanxi
  - Chengdu Fifth People's Hospital, Chengdu, Sichuan
  - Yibin Second People's Hospital, Yibin, Sichuan
  - Yunnan Provincial First People's Hospital, Kunming, Yunnan
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - Jiaxing First Hospital, Jiaxing, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - Beijing Chaoyang Hospital, Beijing
  - Beijing Luhe Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Chongqing jiangjin hospital, Chongqing
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - Inner Mongolia Autonomous Region People's Hospital, Neimeng
  - Chongming Hospital Affiliated to Shanghai University of Medicine & Health Sciences, Shanghai
  - Shanghai Fifth People's Hospital, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - Yichang Central People's Hospital, Yichang

IPD SHARING:
Plan to Share IPD: No